CLINICAL TRIAL: NCT04446403
Title: Analgesic Effect of Ultrasound Guided Combined (Suprascapular and Circumflex Nerve Blocks ) Versus (Suprascapular Nerve and Posterior Cord Nerve Blocks at Infraclavicular Level ) During Shoulder Arthroscopy : A Randomized Controlled Study
Brief Title: Circumflex Nerve Blocks Versus Posterior Cord Nerve Blocks in Shoulder Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bassant M. Abdelhamid (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-10-2019
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- circumflex (Experimental): patients will undergo ultrasound guided SSN+circumflex
  Interventions: Procedure: Suprascapular Nerve Block; Procedure: Axillary Nerve Block; Procedure: General anesthesia
- posterior cord (Experimental): patients will undergo ultrasound guided SSN+circumflex
  Interventions: Procedure: Suprascapular Nerve Block; Procedure: posterior cord block; Procedure: General anesthesia

INTERVENTIONS:
Procedure: Suprascapular Nerve Block — The patient will be put in sitting down position with upper limbs pending beside the body then a high-frequency linear ultrasound probe will be positioned transversely above the spine of the scapula. The suprascapular nerve often appears as hypereccoic structure at the suprascapular notch. A 20-gauge spinal needle will be advanced in-plane from medial to lateral 10mL of bupivacaine 0.25% into the suprascapular notch deep to the superior transverse scapular ligament (STSL) and adjacent to the suprascapular artery (SSA) .
  Other Names: SSN
Procedure: Axillary Nerve Block — Patient will be put in sitting position, with the shoulder in full adduction. linear transducer (8-14 MHz) will be positioned in the short axis orientation at the neck of humerous to identify the axillary artery about 1 to 3 cm from the skin surface.The artery is the most reliable landmark, then a 21-gauge 90 mm needle will be advanced in-plane and 10 mL of bupivacaine 0.25% will be injected adjacent to the artery.
  Arms: circumflex
Procedure: posterior cord block — Patient will be put in supine position with head turned away from side that will be blocked with the arm abducted 90 and flexed at the elbow then linear transducer (8-14 MHz) will be positioned in short-axis just medial to coracoid process.Once the artery will be identified, an attempt will be made to identify the hyperechoic cords of the brachial plexus and their corresponding positions relative to the artery, although these may not always be identifiable. The needle will be inserted in plane from the cephalad end of the probe. 10 mL bupivacaine 0.25% will be injected at the posterior cord.
  Arms: posterior cord
Procedure: General anesthesia — General anaesthesia will be induced after giving nerve block in a standardized way with propofol 1.5-2.5mg/kg, fentanyl 2-3 µ/kg and atracurium 0.5mg/kg. maintenance of anaesthesia with isoflurane and atracurium 0.1mg/kg/20min.

SUMMARY:
Shoulder arthroscopy is associated with severe postoperative pain. Traditionally, the interscalene approach to the brachial plexus has been employed to manage postoperative pain following shoulder surgery.To provide more complete shoulder joint analgesia, suprascabular nerve block (SSNB) was combined with block of the circumflex nerve which comes from the posterior cord of the brachial plexus that usually gives also upper subscapular, thoracodorsal, lower subscapular and radial nerves.

DETAILED DESCRIPTION:
Aim of the work is to compare postoperative analgesic effect of ultrasound guided combined suprascapular and circumflex nerve blocks versus suprascapular nerve and posterior cord blocks at infraclavicular level .

Thirty four patients aged from 18-70 years old, with ASA physical status I-II-III and scheduled for shoulder surgeries will be included in the study. Patients will be randomly allocated using computer-generated table into one of two groups:

* Group circumflex → will undergo ultrasound guided SSN+circumflex.
* Group posterior cord → will undergo ultrasound guided SSN+posterior cord.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II.-III
* Undergoing shoulder arthroscopy.

Exclusion Criteria:

* Patient refusal
* Known allergy to local anesthetics
* Bleeding disorders
* Inability to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Time of the first postoperative analgesic request | 12 hours postoperative

SECONDARY OUTCOMES:
Visual analogue score | 12 hours postoperative
  visual analog scale (VAS) ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain) and verbal pain scale (VPS )ranging from 0 to 3 (0 = no pain, 1 = mild pain, 2 = moderate pain, and 3 = severe pain).
Total morphine consumption | 12 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abd-Elraouf Nasr, Principal Investigator — Cairo University; Ahmed Zaghloul, Study Director — Cairo University; Mohsen Waheb, Study Director — Cairo University
Locations (1):
- Anesthesia Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Axelsson K, Gupta A, Johanzon E, Berg E, Ekback G, Rawal N, Enstrom P, Nordensson U. Intraarticular administration of ketorolac, morphine, and ropivacaine combined with intraarticular patient-controlled regional analgesia for pain relief after shoulder surgery: a randomized, double-blind study. Anesth Analg. 2008 Jan;106(1):328-33, table of contents. doi: 10.1213/01.ane.0000297297.79822.00. PMID 18165599
- [Background] Price DJ. The shoulder block: a new alternative to interscalene brachial plexus blockade for the control of postoperative shoulder pain. Anaesth Intensive Care. 2007 Aug;35(4):575-81. doi: 10.1177/0310057X0703500418. PMID 18020078
- [Background] Lyons C, Herring AA. Ultrasound-guided axillary nerve block for ED incision and drainage of deltoid abscess. Am J Emerg Med. 2017 Jul;35(7):1032.e3-1032.e7. doi: 10.1016/j.ajem.2017.01.064. Epub 2017 Feb 1. PMID 28258838